CLINICAL TRIAL: NCT04835896
Title: An Open Label, Single-arm, Multi-center Phase 1b/2 Combination Study of M7824 (Bintrafusp Alfa) and Paclitaxel in Recurrent/Metastatic Gastric Cancer as a Second-line Treatment
Brief Title: Study of M7824 and Paclitaxel Combination as a Second-line Treatment in Patients With Recurrent/Metastatic Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-1334
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Recurrent/Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental)
  Interventions: Drug: M7824+paclitaxel

INTERVENTIONS:
Drug: M7824+paclitaxel — M7824 will be administered intravenously at a dose of 1200 mg every 3 weeks in combination with paclitaxel 80 (or 70) mg/m2 once a week for 3 weeks (each cycle is 4 weeks)

SUMMARY:
This is a Phase 1b/2 study to identify the recommended dose of M7824 for further study with weekly paclitaxel, and to assess the safety and clinical efficacy of this combined treatment in advanced gastric cancer after first line treatment. The study will be conducted in two parts: Part 1 (Phase 1b) dose escalation study to determine the MTD and RP2D of weekly paclitaxel in combination with fixed dose M7824, Part 2 (Phase 2) to further evaluate the safety and tolerability of the combination of M7824 and paclitaxel at the RP2D and determine anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent and has signed the informed consent form (ICF), prior to performance of any trial activities.
2. Eligible male and female subjects aged ≥19 years.
3. Histologically or cytologically proven metastatic or locally advanced HER2 negative gastric cancer after 1st line failure.
4. ECOG performance status of 0 to 1 at trial entry.
5. Life expectancy ≥12 weeks as judged by the Investigator.
6. Adequate hematological function defined by white blood cell (WBC) count ≥3×109/L with absolute neutrophil count (ANC) ≥1.5×109/L, lymphocyte count ≥0.5×109/L, platelet count ≥100×109/L, and Hb ≥9 g/dL (in absence of blood transfusion).
7. Adequate hepatic function defined by a total bilirubin level ≤1.5×ULN, an AST level ≤1.5×ULN, and an ALT level ≤1.5×ULN. For subjects with liver involvement in their tumor, AST ≤5.0×ULN, ALT ≤5.0×ULN, and bilirubin ≤3.0 is acceptable.
8. Adequate renal function defined by an estimated creatinine clearance >50 mL/min according to the Cockcroft-Gault formula or by measure of creatinine clearance from 24-hour urine collection.
9. Adequate coagulation function: normal international normalized ratio (INR), PT ≤1.5×ULN and activated partial thromboplastin time (aPTT) ≤1.5×ULN.
10. HIV patient must be stable on ART for at least 4 weeks, having documented evidence of multi-drug resistance, viral load of <400 copies/ml and CD4+ T-cells ≤350 cells/µL.
11. HBV/HCV positive participant must be on a stable dose of antiviral therapy, having HBV viral load below the limit of quantification (HBV titer <2000 IU/ml) and HCV RNA is not detected.
12. Has measurable or evaluable disease as determined by RECIST 1.1.

Exclusion Criteria:

1. Concurrent treatment with non-permitted drugs.
2. Prior therapy with any antibody/drug targeting T cell coregulatory proteins (immune checkpoints) such as anti-PD-1, anti-cytotoxic T lymphocyte antigen-4 (CTLA-4) antibody, or anti-4-1BB antibody, is not allowed.
3. Prior therapy with any antibody/drug targeting TGFβ or TGF receptor.
4. Anticancer treatment within 21 days before the start of trial treatment, e.g., cytoreductive therapy, radiotherapy (with the exception of palliative bone-directed radiotherapy), immune therapy, or cytokine therapy.
5. Major surgery within 28 days before the start of trial treatment (excluding prior diagnostic biopsy).
6. Systemic therapy with immunosuppressive agents within 7 days before the start of trial treatment; or use of any investigational drug within 28 days before the start of trial treatment.
7. Has persistent ≥Grade 2 toxicity that was not resolved from previous anticancer treatment, such as neuropathy (exceptions are alopecia and anemia).
8. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation.
9. Has received a live vaccine within 30 days prior to the first dose of study drug.
10. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
11. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years.
12. Has known active CNS metastases and/or carcinomatous meningitis.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
14. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
15. Has an active infection requiring systemic therapy.
16. Has uncontrolled or severe cardiovascular disease, as per following criteria: Myocardial infarction within 180 days before the start of trial treatment; Uncontrolled angina pectoris within 180 days before the start of trial treatment; New York Heart Association (NYHA) Class III or IV congestive heart failure; Uncontrolled hypertension despite appropriate treatment (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg lasting 24 hours or more); Arrhythmia requiring treatment
17. History of bleeding diathesis or recent major bleeding event.
18. Has a known history of Human Immunodeficiency Virus (HIV) without treatment.
19. Has an active of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive and HBV titer >2000 IU/ml) or known active Hepatitis C virus (defined as HCV RNA is detected) infection.
20. Has an active TB (Bacillus Tuberculosis) with treatment.
21. Has known history of hypersensitivity to one or more of the study treatments or their substances, or known severe hypersensitivity to monoclonal antibodies (≥Grade 3), history of anaphylaxis, or uncontrolled asthma within 5 months before start of trial treatment.
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
23. Have received more than 2nd line of chemotherapy.
24. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
25. Otherwise inappropriate for this study in the investigator's or sub-investigator's opinion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Dose-limiting toxicity in subjects with M7824 and paclitaxel combination treatment | Within first 4 weeks
Phase 2: Progression-free survival in subjects with M7824 and paclitaxel combination treatment | At 24 weeks

SECONDARY OUTCOMES:
Overall survival | 3 months after the last dose study treatment of the last subject
Objective response rate according to RECIST 1.1 | 3 months after the last dose study treatment of the last subject
Disease control rate according to RECIST 1.1 | 3 months after the last dose study treatment of the last subject
Duration of response according to RECIST 1.1 | 3 months after the last dose study treatment of the last subject
Progression-free survival according to RECIST 1.1 | 3 months after the last dose study treatment of the last subject
Safety and Tolerability, in terms of the number, severity, and duration of treatment-emergent adverse events as assessed by CTCAE v5.0 | Throughout the overall trial period as well as up to 3 months after the last dose study treatment for each subject

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young RHA, MD, PhD, Principal Investigator — Yonsei Cancer Center, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No